CLINICAL TRIAL: NCT03986866
Title: Video-based, Patient-Focused Opioid Education in the Perioperative Period: A Feasibility Study
Brief Title: Video-based, Patient-Focused Opioid Education in the Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 228789
Record Dates: First submitted 2019-06-05; First posted 2019-06-14 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2021-12

CONDITIONS: Opioid Use; Chronic Pain Post-Procedural
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Video (No Intervention): Patients are not shown the informational video on the safe usage of opioids.
- Video (Experimental): Patients are shown an informational video on the safe usage of opioids.
  Interventions: Other: Video

INTERVENTIONS:
Other: Video — A 5 minute video on the risks and benefits of opioids, alternative methods to reduce pain, and the proper handling and storage of opioids will be shown.
  Arms: Video

SUMMARY:
This is a pilot study designed to assess the feasibility of using a novel, video-based opioid education tool for opioid naïve ambulatory surgery patients in the perioperative period.

DETAILED DESCRIPTION:
Patients will be randomized to a video or no video prior to surgery then administered a phone questionnaire at post-op day 7, 30, and 90. The Arkansas Prescriptions Drug Monitoring Database will also be accessed for information on opioid prescription refills. The overall goal of the study is to evaluate the effect that video-based opioid education has on narcotic intake after outpatient surgery. The duration of the study will be approximately 3 months, plus a single 1-hour long focus group if desired by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years or older
* Not chronically receiving opioid analgesics
* Patients who have not taken opioids 30 days pre-operatively
* Undergoing surgical procedure not requiring overnight hospital stay

Exclusion Criteria:

* Non-English speaking
* Legally deaf or blind
* On opiate contract
* Has taken oral narcotic in the past 30 days
* Unable to operate a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan H Goree, M.D., Principal Investigator — University of Arkansas; Lauren Byers, APRN, Study Chair — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Ayasrah SM, Ahmad MM. Educational Video Intervention Effects on Periprocedural Anxiety Levels Among Cardiac Catheterization Patients: A Randomized Clinical Trial. Res Theory Nurs Pract. 2016;30(1):70-84. doi: 10.1891/1541-6577.30.1.70. PMID 27025001
- [Background] Basch CE. Focus group interview: an underutilized research technique for improving theory and practice in health education. Health Educ Q. 1987 Winter;14(4):411-48. doi: 10.1177/109019818701400404. PMID 3319971
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Chakravarthy B, Somasundaram S, Mogi J, Burns R, Hoonpongsimanont W, Wiechmann W, Lotfipour S. Randomized pilot trial measuring knowledge acquisition of opioid education in emergency department patients using a novel media platform. Subst Abus. 2018 Jan 2;39(1):27-31. doi: 10.1080/08897077.2017.1375061. Epub 2017 Sep 29. PMID 28873050
- [Background] Deyo RA, Hallvik SE, Hildebran C, Marino M, Dexter E, Irvine JM, O'Kane N, Van Otterloo J, Wright DA, Leichtling G, Millet LM. Association Between Initial Opioid Prescribing Patterns and Subsequent Long-Term Use Among Opioid-Naive Patients: A Statewide Retrospective Cohort Study. J Gen Intern Med. 2017 Jan;32(1):21-27. doi: 10.1007/s11606-016-3810-3. Epub 2016 Aug 2. PMID 27484682
- [Background] Hill AM, McPhail S, Hoffmann T, Hill K, Oliver D, Beer C, Brauer S, Haines TP. A randomized trial comparing digital video disc with written delivery of falls prevention education for older patients in hospital. J Am Geriatr Soc. 2009 Aug;57(8):1458-63. doi: 10.1111/j.1532-5415.2009.02346.x. Epub 2009 Jun 8. PMID 19515102
- [Background] Krebs EE, Gravely A, Nugent S, Jensen AC, DeRonne B, Goldsmith ES, Kroenke K, Bair MJ, Noorbaloochi S. Effect of Opioid vs Nonopioid Medications on Pain-Related Function in Patients With Chronic Back Pain or Hip or Knee Osteoarthritis Pain: The SPACE Randomized Clinical Trial. JAMA. 2018 Mar 6;319(9):872-882. doi: 10.1001/jama.2018.0899. PMID 29509867
- [Background] Meissner W, Coluzzi F, Fletcher D, Huygen F, Morlion B, Neugebauer E, Montes A, Pergolizzi J. Improving the management of post-operative acute pain: priorities for change. Curr Med Res Opin. 2015 Nov;31(11):2131-43. doi: 10.1185/03007995.2015.1092122. Epub 2015 Sep 30. PMID 26359332
- [Background] Memtsoudis SG, Poeran J, Zubizarreta N, Cozowicz C, Morwald EE, Mariano ER, Mazumdar M. Association of Multimodal Pain Management Strategies with Perioperative Outcomes and Resource Utilization: A Population-based Study. Anesthesiology. 2018 May;128(5):891-902. doi: 10.1097/ALN.0000000000002132. PMID 29498951
- [Background] Oliver JW, Kravitz RL, Kaplan SH, Meyers FJ. Individualized patient education and coaching to improve pain control among cancer outpatients. J Clin Oncol. 2001 Apr 15;19(8):2206-12. doi: 10.1200/JCO.2001.19.8.2206. PMID 11304773
- [Background] Pereira L, Figueiredo-Braga M, Carvalho IP. Preoperative anxiety in ambulatory surgery: The impact of an empathic patient-centered approach on psychological and clinical outcomes. Patient Educ Couns. 2016 May;99(5):733-8. doi: 10.1016/j.pec.2015.11.016. Epub 2015 Nov 26. PMID 26654958
- [Background] Prabhu M, Dubois H, James K, Leffert LR, Riley LE, Bateman BT, Henderson M. Implementation of a Quality Improvement Initiative to Decrease Opioid Prescribing After Cesarean Delivery. Obstet Gynecol. 2018 Sep;132(3):631-636. doi: 10.1097/AOG.0000000000002789. PMID 30095765
- [Background] Sabatino MJ, Kunkel ST, Ramkumar DB, Keeney BJ, Jevsevar DS. Excess Opioid Medication and Variation in Prescribing Patterns Following Common Orthopaedic Procedures. J Bone Joint Surg Am. 2018 Feb 7;100(3):180-188. doi: 10.2106/JBJS.17.00672. PMID 29406338
- [Background] Safeer RS, Keenan J. Health literacy: the gap between physicians and patients. Am Fam Physician. 2005 Aug 1;72(3):463-8. PMID 16100861
- [Background] Shah A, Hayes CJ, Martin BC. Characteristics of Initial Prescription Episodes and Likelihood of Long-Term Opioid Use - United States, 2006-2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 17;66(10):265-269. doi: 10.15585/mmwr.mm6610a1. PMID 28301454
- [Background] Sobo EJ, Seid M, Reyes Gelhard L. Parent-identified barriers to pediatric health care: a process-oriented model. Health Serv Res. 2006 Feb;41(1):148-72. doi: 10.1111/j.1475-6773.2005.00455.x. PMID 16430605
- [Background] Theisen KM, Myrga JM, Hale N, Cochran G, Sewall C, Macleod LC, Jacobs BL, Davies BJ. Excessive Opioid Prescribing After Major Urologic Procedures. Urology. 2019 Jan;123:101-107. doi: 10.1016/j.urology.2018.06.057. Epub 2018 Aug 24. PMID 30149041
- [Background] Thiels CA, Hanson KT, Cima RR, Habermann EB. From Data to Practice: Increasing Awareness of Opioid Prescribing Data Changes Practice. Ann Surg. 2018 Mar;267(3):e46-e47. doi: 10.1097/SLA.0000000000002623. PMID 29215369
- [Background] Valentine AR, Carvalho B, Lazo TA, Riley ET. Scheduled acetaminophen with as-needed opioids compared to as-needed acetaminophen plus opioids for post-cesarean pain management. Int J Obstet Anesth. 2015 Aug;24(3):210-6. doi: 10.1016/j.ijoa.2015.03.006. Epub 2015 Mar 23. PMID 25936786
- [Background] Watt-Watson J, Stevens B, Costello J, Katz J, Reid G. Impact of preoperative education on pain management outcomes after coronary artery bypass graft surgery: a pilot. Can J Nurs Res. 2000 Mar;31(4):41-56. PMID 11189670
- See also: Publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8403019/pdf/jpr-14-2583.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Video | Video
Started | 55 | 55
Completed | 53 | 50
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 0 | 3
Not completed — patient required admission so no longer fit study exclusion criteria of ambulatory surgery | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patients who after randomization have an outpatient surgical encounter
Groups:
- Total: Total of all reporting groups
Arm/Group | No Video | Video | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 39 | 85
  >=65 years | 7 | 11 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 24 | 16 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Knowledge of Post Operative Opioids
Description: Knowledge of Post operative Opioids after surgery via 7 day post operative phone call. Knowledge is measured on a scale of 1 to 10 with 10 being complete knowledge and 1 being no knowledge.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Video | Video
Number analyzed (Participants) | 36 | 33
units on a scale | 8.32 (2.5) | 9.36 (1.2)

2. Primary Outcome: Number of Patients Who Discontinued Opioids by 3 Months
Description: Post-operative pain control as determined by opioid utilization at three months. This is the number of patients that have discontinued opioids at the 3 month mark.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | No Video | Video
Number analyzed (Participants) | 53 | 50
Participants | 47 | 38

3. Secondary Outcome: Development of Chronic Opioid Use
Description: Feasibility of collecting data on the percentage of patients who develop chronic opioid use. This is measured as the number of patients who received an opioid prescription per the Arkansas prescription drug monitoring database during the 90-150 day period post operatively.
Time Frame: 90-150 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Video | Video
Number analyzed (Participants) | 53 | 50
Participants | 12 | 5

4. Secondary Outcome: Number of Total Days to Opioid Cessation
Description: Feasibility of collecting data on the number of days until opioid cessation
Time Frame: Up to 3 months
Population: Days until opioid cessation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | No Video | Video
Number analyzed (Participants) | 30 | 29
days | 13.9 (17) | 13.9 (20.9)

ADVERSE EVENTS:
Time Frame: three months post enrollment
Arm/Group | No Video | Video
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 0/53 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT03986866/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT03986866/ICF_001.pdf